CLINICAL TRIAL: NCT04810312
Title: Combined Exercise and Nutrition Intervention for Spinal Sarcopenia: a Pilot Study
Brief Title: Combined Exercise and Nutrition Intervention for Spinal Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Yoon Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-2021-27
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia
Keywords: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Back extensor strengthening with oral protein supplementation
  Interventions: Other: Combined exercise and nutrition intervention

INTERVENTIONS:
Other: Combined exercise and nutrition intervention — Back extensor strengthening exercise and nutritional supplementation for 12 weeks

SUMMARY:
Sarcopenia in the lumbar paraspinal muscles is receiving renewed attention as a cause of spinal degeneration. However, there were few studies on the precise concept and diagnostic criteria for spinal sarcopenia. We have already developed the concept of spinal sarcopenia in community-dwelling older adults and investigated the association between conventional sarcopenic indices and spinal sarcopenia. However, intervention studies on spinal sarcopenia have not been conducted until now. Here, we aim a pilot study to evaluate the effectiveness of the combined exercise and nutrition intervention for spinal sarcopenia.

This is a prospective study with 35 community-dwelling older women who were diagnosed as spinal sarcopenia in our previous cohort study. Combined intervention will consist of back extensor strengthening exercise and nutritional supplementation for 12 weeks. The primary outcome of this study is isometric back extensor strength after 12 weeks' intervention. All functional outcomes will be measured at 0, 12, and 24 weeks after intervention. The data will be analysed using the intention-to-treat principle.

DETAILED DESCRIPTION:
Both the atrophy and fatty change of paraspinal muscles originated from sarcopenia on lumbar paraspinal are also known to be associated with functional disorders and chronic back pain. We want to suggest classifying this phenomenon as "spinal sarcopenia." While feasible, inexpensive, and less radiation-exposed tools such as dual energy X-ray absorptiometry have been used to measure appendicular skeletal muscle mass, paraspinal muscle assessment is still needed using spinal CT or MRI. In addition, spinal extensor strength measurement is necessary to confirm the function of lumbar paraspinal muscle, but isokinetic exercise equipment for accurate measurement is not as feasible as a dynamometer for hand grip strength to evaluate sarcopenia. Furthermore, many elderly people may experience pain during the measurement of spinal extension strength. Therefore, it is necessary to develop a simple, accessible, and clinically meaningful measurement index to confirm the myofunction of spinal extension. The main two axes of treatment and prevention of conventional sarcopenia are muscle strengthening exercises and high protein nutritional supplements. Therefore, it is necessary to confirm the clinical effect by intervention for spinal extension exercise and nutritional supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Older women (≥ 65 years old)
* Community-dwellers
* Able to walk with or without assistive devices for more than 100 meters

Exclusion Criteria:

* Low back pain with moderate severity (numeric rating scale 5 and over)
* History of any types of lumbar spine surgery
* History of hip fracture surgery and arthroplasty of hip or knee
* Contraindications for MRI (such as cardiac pacemaker, implanted metallic objects, and claustrophobia)
* Disorders in central nervous system (such as stroke, parkinsonism, spinal cord injury)
* Cognitive dysfunction (Mini Mental State Examination score < 24)
* Communication disorder (such as severe hearing loss)
* Musculoskeletal condition affecting physical function (such as amputation of limb)
* Long-term use of corticosteroids due to inflammatory disease
* Malignancy requiring treatment within 5 years
* Other medical conditions which need active treatment
* Subjects who refuse to participate in a study

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Isometric back extensor strength | 12 weeks after intervention
  Isometric back muscle strength test using a handheld dynamometer (PowerTrack II; JTECH Medical, Salt Lake City, UT, USA)

SECONDARY OUTCOMES:
Isometric back extensor strength | 24 weeks after intervention
  Isometric back muscle strength test using a handheld dynamometer Shirley, NY, USA) to measure the torque of the back extensors
Isokinetic back extensor strength | 12 weeks after intervention
  Isokinetic dynamometer (Biodex multi-joint system, Biodex Corporation, Shirley, NY, USA) to measure the torque of the back extensors
Isokinetic back extensor strength | 24 weeks after intervention
  Isokinetic dynamometer (Biodex multi-joint system, Biodex Corporation, Shirley, NY, USA) to measure the torque of the back extensors
Lumbar paraspinal muscle volume | 12 weeks after intervention
  Lumbar spine MRI will be performed using a 1.5-T scanner (Achieva 1.5 T; Philips Healthcare, Netherlands)
Short physical performance battery (SPPB) | 12 weeks after intervention
  Physical performance test (0-12)
Short physical performance battery (SPPB) | 24 weeks after intervention
  Physical performance test (0-12)
Spinal sagittal balance parameters | 12 weeks after intervention
  Sagittal vertical axis (SVA) distance (mm)
Spinal sagittal balance parameters | 24 weeks after intervention
  Sagittal vertical axis (SVA) distance (mm)

CONTACTS AND LOCATIONS:
Overall Officials: SANG YOON LEE, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center